CLINICAL TRIAL: NCT07080203
Title: Effects of Uterine Prolapse Symptoms Based on Degrees and Their Relation to Quality of Life in the Childbearing Period
Brief Title: Quality of Life Assessment in Patients With Different Degrees of Pelvic Organ Prolapse
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hatem Awaga, Assistant professor, Sohag University
Other Study IDs: Soh-Med-23-12-04MS
Record Dates: First submitted 2025-07-14; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Degree of Uterine Prolapse and Its Effect on Quality of Life
Keywords: Uterine Prolapse; Quality of Life; Childbearing period
MeSH Terms: conditions — Uterine Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- group 1: all available women attending outpatient clinics at sohag university hospital and according to the pilot study and demand of the women to clinical investigations also authenticity for the P-QOL. Questionnaire the Quasi experimental research design with purposive sample from the convenient sample were used to confirm the diagnosis and make intervention to improve the quality of life for that women.

SUMMARY:
Study design:

The study building by two design a descriptive exploratory research design and quasi experimental research design were utilized in the present study

Setting of the study:

This study was conducted at the Outpatient Clinics of Sohag university hospital after approval from the Sohag university medical ethics committee and nursing ethics committee.

Subjects of the study

Sampling:

the sample consists of 400 women.

Sample technique:

a convenient sample of all available women attending outpatient clinics at sohag university hospital and according to the pilot study and demand of the women to clinical investigations also authenticity for the P-QOL. Questionnaire the Quasi experimental research design with purposive sample from the convenient sample were used to confirm the diagnosis and make intervention to improve the quality of life for that women .

Tools of study:

Two tools were utilized and filled by researchers for collecting the data of this study.

The First Tool:

Structured interviewing questionnaire developed by the researcher based on relevant literature divided into three parts.

Part I: socio demographic data as; (age, level of education , income , marital status , place of residence, occupation,).

Part II: Medical history: Related to chronic constipation ,chronic cough and other chronic diseases.

Part III: obstetrical history: Includes (number of pregnancies, number of vaginal deliveries, inter pregnancy interval)

The second Tool: P-QOL. questionnaire adopted from (Digesu et al., 2005) and consist of 9 items (General health perceptions, Prolapse impact, Role limitations, Physical limitations, Social limitations, Personal relationships, Emotions, sleep /energy , Severity measures) then after detect and to determine the degree of prolapse were referred to gynecological clinic to be investigated by clinical supervisor.

Scoring system:

The researcher collected data from patients to complete the P-QOL questionnaire to assess how much their symptoms (if present) were affecting them. Responses ranged from ''not at all, through ''slightly'', ''moderately'' to ''a lot'', from very good to very poor and never to all the time. Therefore, a four- or five-point scoring system according each item was used for severity measurement of uterine prolapse symptoms. Scores in each domain range between 0 and 100. A high total score indicates a greater impairment of quality of life, while a low total score indicates a good quality of life.

* A score from 0 to 50 indicates women has good quality of life with no symptoms of uterine prolapse
* A score more than 50 indicates women has impairment of quality of life and need to clinical evaluation to confirm the degree with symptoms of uterine prolapse.

Tool Validity and Reliability:

Validity:

The validity was assessed by measuring levels of missing data, comparing symptom scores between affected and asymptomatic women and lastly comparing symptom scores with objective vaginal examination related to stages of uterine prolapse, in the symptomatic group, as described in the POP-Q, using Spearman's correlation coefficient (construct validity). (Digesu et al., 2005).

Reliability:

The reliability of the questionnaire was assessed by its internal consistency using the Cronbach alpha and stability using a 2-week test-retest analysis. Internal consistency refers to the degree of correlation between the items. Therefore, it is expected that items forming a domain should moderately correlate with each other, but should contribute independently to the overall domain score. A perfect correlation of 1.0 indicates that the questions are measuring an identical construct. A poor correlation instead suggests that the items are testing different traits. A Cronbach alpha of >0.7 has been recommended as acceptable. (Digesu et al., 2005).

Pilot study:

It was carried out on 40 women to understand the feasibility of participant recruitment regarding study design and to ensure that the respondents for the pilot should be as similar as possible for the actual items in terms of age, gender, education, socioeconomic (income) status. It also helped in the estimation of the time needed to fill the tool .Women who participated in pilot study were included in the main study because because no modifications needed to be performed and five cases of them have uterine prolapse symptoms need clinical examination.

DETAILED DESCRIPTION:
* Preparatory phase It included reviewing past, current, local and international related literature and theoretical knowledge of various aspects of the study using books, articles, internet, periodicals and magazines regarding of the effects of uterine prolapse symptoms based on degrees and their relation to quality of life in the childbearing period . the researcher attended the previously mentioned setting twice or sometimes three times per week from 8 Am to 12 p.m .
* First step The researcher obtained approval from the dean of the Faculty of Nursing at Sohag University, Dean of the Faculty of Medicine at sohag university and director of sohag university hospital
* Second step The researcher met with all the women in the childbearing period convenient in outpatient clinics twice weekly and sometimes three times per week after the researcher introduced herself, explained the goal of the study to them , and obtained formal consent from each women who agreed to participate in the study. Confidentiality of any information obtained was guaranteed, and subjects were informed of their right to participate or not to participate in the study. Anonymity is also assured, and this data will only be used for the study.

Data was collected and filled by the researcher via interviewing questionnaire at the beginning the women were asked about their sociodemographic data and medical and obstetric history then they were asked on items included in P-QOL questionnaire which was adopted from (Digesu et al., 2005) and consists of 9 items (General health perceptions which include questions such (How would you describe your health at present and How much do you think your prolapse problem affect your life) , Prolapse impact which include urinary and vaginal symptoms such (Going to the toilet to pass urine very often, Urgency:A strong desire to pass urine, Urge incontinence ; urinary leakage associated with a strong desire to pass urine, Stress incontinence ; urinary leakage associated with coughing, Feeling a bulge / lump from or in the vagina , Heaviness or dragging feeling as the day goes on from the vagina or the lower abdomen, Vaginal bulge interfering with you emptying your bowels, Discomfort in the vagina which is worse when standing and relieved by lying down, Poor urinary stream, straining to empty your bladder and Urine dribbles after emptying your bladder) ,bowel and vaginal symptoms which include (Bowels do not feel completely empty after opening, Constipation ;difficulty in emptying, Straining to open your bowels, vaginal bulge which gets in the way of sex, Lower backache worsens with vaginal discomfort, Do you help empty your bowels with your fingers? How often do you open your bowels? , Role limitation which include questions such as ( To what extent does your prolapse affect your household tasks ( e.g. cleaning ,shopping )? And Does you prolapse affect your job or your normal daily activities outside the home ?) , Physical and social limitations which include questions such as (Does your prolapse affect your physical activities (e.g. going for a walk , run , sport , gym etc.)?, Does your prolapse affect your ability to travel, Does your prolapse limit your social life? And Does your prolapse limit your ability to see/visit friends ?) , Personal relationships which include such as(Does your prolapse affect your relationship with your partner ?, Does your prolapse affect your sex life? and Does your prolapse affect your family life?.) , Emotions which include questions such as ( Does your prolapse make you feel depressed, Does your prolapse make you feel anxious or nervous ? and Does your prolapse make you feel bad about you self?) , sleep /energy questions which include (Does your prolapse affect your sleep ?and Do you feel worn out / tired ?) ,Severity measures which include(Use tampons /pads /firm knickers to help?, Do you push up the prolapse?, Pain or discomfort due to the prolapse ? and Does the prolapse prevent you from standing ?).

After the women answered these questions. According to the reported symptoms by the women the researcher knew if the women have symptoms of uterine prolapse or no and have good quality of life or impairment in quality of life according to scoring system in P-QOL questionnaire . Once the questionnaires had been completed and collected, an explanation of what had been measured was given to the women and assurances were given also and the women with uterine prolapse symptoms and have impairment of quality of life were told that they need to clinical examination to confirm if they have uterine prolapse or no and if they have uterine prolapse which degree they have. Moreover the researcher explained by booklet for the women about uterine prolapse definition ,causes, risk factors, degrees, symptoms and how to prevent themselves from having uterine prolapse Then the researcher told the women having uterine prolapse symptoms to be in contact with her to find near available time with the physician for clinical examination .

-Third step The researcher was in contact with the physician to determine an available time to examine cases which have symptoms of uterine prolapse . and then the researcher told the women through their mobile phone about time for examination determined by physician .that was about three times monthly every time about four or five cases according to accessibility came for clinical examination .Examination for cases occurred in two places in Feto-maternal unit in special clinics and department of obstetric and gynecology (OBGYN) in sonography room . when the women arrived to hospital waiting room during this the researcher repeated what had been explained for the women about uterine prolapse definition ,causes, risk factors, degrees, symptoms and how to prevent themselves from having uterine prolapse after that the women came to the examination room which was prepared before women coming with sterile Cusco-speculum according to number of cases and sterilization of examination bed then women are asked to empty her bladder before entering the room then women entered the room and nurse in examination room asked the women to keep her clothes down and put women in supine position with knee slightly flexed and rotated outward with complete keeping privacy during examination . after that physician wear gloves and begin to examine cases per vaginal examination at first uses transvaginal sonography to screen uterus ,ovaries ,fallopian tube ,endometrium for any lesion ,polyp, cyst and myoma then sterile Cusco-speculum with lubricated gel slightly inserted through the vagina to determine uterine decent especially in cases of first degree uterine prolapse where cannot be seen through the vaginal decent because in first degree uterine prolapse cervix is below ischial spine then prevaginal examination is done and physician put his fingers in posterior wall of the vagina and ask women to cough to see if there is any vaginal bulge this help to determine if women have cystocele or no and repeat this in anterior wall of the vagina to detect if women has rectocele or no. then physician removed gloves and ask women to be in comfortable position . with examination physician detected some problems which women have as urinary tract infection such as vaginitis or cervicitis so physician described proper treatment for such cases as well as told and reassure women how to manage uterine prolapse according to degree and the researcher repeated what physician has said to women and help in direction of cases to follow physician instructions Lastly, after finishing lots of thanks were given to women for their cooperation.

There were about 50 women which don't have any uterine prolapse symptoms asked if they allowed to do clinical examination to confirm that if they have uterine prolapse or no so clinical examination was done for them and illustrated that they actually don't have uterine prolapse .

Administrative design:

An official letter approval was obtained from Dean of the Faculty of Medicine and Faculty of Nursing at Sohag University to directors of previous setting in Sohag University. This letter included a brief explanation of the objectives of the study and permission to carry out the study

ELIGIBILITY:
Inclusion Criteria:

women in the childbearing period convenient in outpatient clinics twice weekly and sometimes three times per week

Exclusion Criteria:

-

Min Age: 18 Months | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — only females are expected to have prolapse and eligible for the current study
Study Population: The researcher met with all the women in the childbearing period convenient in outpatient clinics twice weekly and after the researcher introduced herself, explained the goal of the study to them , and obtained formal consent from each women who agreed to participate in the study. Confidentiality of any information obtained was guaranteed, and subjects were informed of their right to participate or not to participate in the study. Anonymity is also assured, and this data will only be used for the study. Data was collected and filled by the researcher via interviewing questionnaire at the beginning the women were asked about their sociodemographic data and medical and obstetric history then they were asked on items included in P-QOL questionnaire which was adopted from (Digesu et al., 2005).and the women with uterine prolapse symptoms and have impairment of quality of life were told that they need to clinical examination to assess the degree of uterine prolapse.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
effect of uterine prolapse on quality of life | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
decision is still under discussion by all research team

REFERENCES:
- [Background] Tega A, Yenealem F, Belay G, Asmare E, Getaneh T, Desalegn M, Dechasa N, Addis Z. Quality of life and its associated factors among women with pelvic organ prolapse who attend gynecology clinics Southern Ethiopia 2022. BMC Womens Health. 2024 Jul 12;24(1):398. doi: 10.1186/s12905-024-03238-1. PMID 38997642
- [Background] Tefera Z, Temesgen B, Arega M, Getaneh T, Belay A. Quality of life and its associated factors among women diagnosed with pelvic organ prolapse in Gynecology outpatient department Southern Nations, Nationalities, and Peoples region public referral hospitals, Ethiopia. BMC Womens Health. 2023 Jun 28;23(1):342. doi: 10.1186/s12905-023-02507-9. PMID 37380942
- [Background] Tahmina Afrin ., Furatul,H., Shahidul,I., Zahid ,B., Zakia ,R., Abid ,H., Abul Kasem ,M.( 2017-2018) DU Roll: 1292 Reg no: 10223, Quality of Life Among women Having Genital Prolapse, Saic College of Medical Science and Technology Department of physiotherapy )
- [Background] Shehata Ibrahim, S., Mohamed Elbhlwan, G. A., & Mansour, S. A. (2023). Knowledge and Practices of Women Regarding Risk Factors and Preventive Measures of Vaginal Prolapse. Port Said Scientific Journal of Nursing, 10(2), 299-319.
- [Background] Rashad, M., Fadel, E., & El-Nemer, A. (2018). Women's knowledge regarding pelvic organ Shavkatovich, S. X. (2025). Incidence Rates of Genital Prolapse in Women of Reproductive Age. Web of Medicine: Journal of Medicine, Practice and Nursing, 3(1), 145-149.
- [Background] Ramadan Hassan, S. G., Moustafa, M. F., Mohamed, H. A. E., El-Malek, A., & Samier, A. (2020). Effect of Kegel Exercise on Improving Manifestations of Uterine Prolapse among Pre menopausal Women. Minia Scientific Nursing Journal, 8(1), 75-82.
- [Background] Olimjonovna, T. D. (2025). UTERINE PROLAPSE IS A DELICATE PROBLEM FOR WOMEN. Modern education and development, 19(3), 163-171. prolapse. Mansoura Nursing Journal, 5(3), 57-67.
- [Background] Okonofua, F., Balogun, J. A., Odunsi, K., & Chilaka, V. N. (Eds.). (2021). Contemporary obstetrics and gynecology for developing countries. Springer.
- [Background] Mohammed Saeed, N., Mohamed Fahmy, N., Abdelhalem Said, S., & Abozied Ramadan, E. (2022). Effect of Nursing Intervention Package on Prevention of Uterine Prolapse among Pregnant Women in Third Trimester. Journal of Nursing Science Benha University, 3(1), 918-939.
- [Background] Martins, F. E. (2025). Pelvic Organ Prolapse and Sexual Dysfunction. Société Internationale d'Urologie Journal, 6(1), 19.
- [Background] Kurniadi A, Dewi AK, Sasotya RMS, Purwara BH, Kireina J. Effect of Vitamin D analog supplementation on levator ani strength and plasma Vitamin D receptor expression in uterine prolapse patients. Sci Rep. 2023 Mar 3;13(1):3616. doi: 10.1038/s41598-023-30842-2. PMID 36869168
- [Background] Kayondo M, Kaye DK, Migisha R, Tugume R, Kato PK, Lugobe HM, Geissbuehler V. Impact of surgery on quality of life of Ugandan women with symptomatic pelvic organ prolapse: a prospective cohort study. BMC Womens Health. 2021 Jun 25;21(1):258. doi: 10.1186/s12905-021-01397-z. PMID 34172043
- [Background] K Khalil, A., Ahmed Mohmed Elbahlowan, G., E Nady, S., & ES, A. (2024). Guidelines for Nursing Care: Effect on Quality of Sexual Life among Women with Vaginal Prolapse. Egyptian Journal of Health Care, 15(4), 818-832.
- [Background] Jayashree, K., Indira, A., & Viji, A. (2022). Impact Of Nurse Led Bundle Care Therapy On Pop Symptoms Among Women With Prolapsed Uterus. Journal of Pharmaceutical Negative Results, 125-131.
- [Background] Gonzalez-Timoneda A, Valles-Murcia N, Munoz Esteban P, Torres Lopez MS, Turrion Martinez E, Errandonea Garcia P, Serrano Raya L, Nohales Alfonso F. Prevalence and impact of pelvic floor dysfunctions on quality of life in women 5-10 years after their first vaginal or caesarian delivery. Heliyon. 2025 Jan 21;11(3):e42018. doi: 10.1016/j.heliyon.2025.e42018. eCollection 2025 Feb 15. PMID 39916837
- [Background] Gomathi, K., Mazumder, S., Soniya, M., & Jenifer, S. (2020). A study to assess the knowledge on uterine prolapse among reproductive age group women's in Kudamoakkam. Int J Midwifery Nurs Pract, 3(2), 11-13. www.nursingpractice.net.
- [Background] Fathi Mohammed, R., D Mohammed, M., & Hassan Abd El-Rahim, A. (2021). Determinants and Symptoms Severity of Pelvic Organ Prolapse and Its Effect on Physical Activities among the Elderly versus Childbearing Women. Egyptian Journal of Health Care, 12(1), 664-685. Giri, S. (2023).
- [Background] Elsayed1F, Ahmed M, Sayed M, Gaheen A (2016). Knowledge and Practices of women regarding Risk Factors of Uterine Prolapse, Ahmed Uterine Prolapse Treatment & Management. IOSR Journal of Nursing and Health Science (IOSR-JNHS)e-ISSN: 2320- 1959.p- ISSN: 2320-1940 Volume 5, Issue 6 Ver. III (Nov. - Dec. 2016), PP 60 67www.iosrjournals.orgDOI:10.9790/1959050 6036067www.iosrjournals.org60Page Updated: Mar 05, 2020
- [Background] El Kady O, Tamara T, Abd ElMohsen H., & Mohamed A. (2017). Assessment of The Prevalence of Pelvic Floor Disorders in Both Vaginal and Cesarean Deliveries and Their Impact on The Quality of Life. The Egyptian Journal of Hospital Medicine.Vol.68 (2), Page 12521256.
- [Background] Eid Abd El-Hamid, N., Ahmed Hassan Omran, A., Ibrahim, A. E. H. S., & Amin Ali Gafar, H. (2023). Assessment of Womens Knowledge, Practices and Attitudes regarding Uterine Prolapse. Journal of Nursing Science Benha University, 4(1), 191-203.
- [Background] Devkota HR, Sijali TR, Harris C, Ghimire DJ, Prata N, Bates MN. Bio-mechanical risk factors for uterine prolapse among women living in the hills of west Nepal: A case-control study. Womens Health (Lond). 2020 Jan-Dec;16:1745506519895175. doi: 10.1177/1745506519895175. PMID 31965915
- [Background] Bogati, N. K., Aryal, B., Kuikel, J., Bogati, T., & Ranabhat, C. L. (2023). Prevalence and Risk Factors of Uterine Prolapse in Achham District, Nepal. Journal of Health Promotion, 11(1), 32-47. DOI: 10.3126/jhp.v11i1.61200
- [Background] Belayneh T, Gebeyehu A, Adefris M, Rortveit G, Gjerde JL, Ayele TA. Pelvic organ prolapse surgery and health-related quality of life: a follow-up study. BMC Womens Health. 2021 Jan 2;21(1):4. doi: 10.1186/s12905-020-01146-8. PMID 33388056
- [Background] Badacho AS, Lelu MA, Gelan Z, Woltamo DD. Uterine prolapse and associated factors among reproductive-age women in south-west Ethiopia: A community-based cross-sectional study. PLoS One. 2022 Jan 21;17(1):e0262077. doi: 10.1371/journal.pone.0262077. eCollection 2022. PMID 35061761
- [Background] Addisu D, Mekie M, Belachew YY, Degu A, Gebeyehu NA. The prevalence of pelvic organ prolapse and associated factors in Ethiopia: a systematic review and meta-analysis. Front Med (Lausanne). 2023 Jul 5;10:1193069. doi: 10.3389/fmed.2023.1193069. eCollection 2023. PMID 37476611